CLINICAL TRIAL: NCT01655654
Title: Prevalence, Awareness and Management of Hypertension in Acute Care Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSWR-002-EHW
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: Hypertension; Acute hospital staff; Exercise; Diet
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (No Intervention): All employees within the acute care hospital that signed the informed consent form and provided their individual data.
- Cohort 2 (Active Comparator): All subjects of cohort 1 who also are considered hypertensive and participated in one or more study interventions, which include behavioral interventions (an increase in physical activity, or dietary changes) or who have a primary care provider visit to discuss hypertension.
  Interventions: Behavioral: Physical activity; Behavioral: Dietary; Other: Primary care provider visit

INTERVENTIONS:
Behavioral: Physical activity — This intervention includes cardiorespiratory exercise, resistance exercise, flexibility exercise and neuromotor exercise.
  Arms: Cohort 2
Behavioral: Dietary — Make at least one positive dietary change including or similar to a DASH diet snack substitution.
  Arms: Cohort 2
Other: Primary care provider visit — Subjects with hypertension will be asked to visit their primary care provider seeking treatment options. If a subject does not have a primary care provider then they will be encouraged to obtain one and seek medical treatment.
  Arms: Cohort 2

SUMMARY:
The primary purpose of this study is to identify the percentage of health care workers working in an acute care hospital who have high blood pressure, to determine the awareness of their blood pressure status, and to see how well it is managed. Study participants will come from the following three distinctly different types of departments: telemetry (clinical), non-telemetry (clinical), and non-direct patient care staff. All study participants are offered educational information surrounding high blood pressure and review the recommendation for their primary care engagement. Study participants with high blood pressure will be asked to continue in the study for up to 6 months. It is intended that each study participant who continues will take their blood pressure three times a day and record the results in a study provided diary. Each study participant should also make some of the suggested changes that promote a healthier lifestyle including exercising, improving their diet, and seeing their primary care provider. It is the thought that these changes will reduce the study participant's blood pressure. The secondary purpose is to determine the effect shift work has on these hospital employees and the potential positive effects of the three interventions.

DETAILED DESCRIPTION:
Research on hypertension (HTN) in hospital personnel during work hours is limited yet research has been published on the relationship of job strain and the risk of cardiovascular disease. HTN can be caused by sympathoadrenal activation brought on by long-term exposure to stressors and an inherent biomarker that is associated with an increased risk of cardiovascular disease.

The primary purpose of this study is to quantify differences in HTN prevalence, awareness and management in three distinctly different areas and shifts within an acute hospital. Blood pressure (BP) will be taken during working hours along with pre and post sleep hours. The secondary purpose is to identify the effect of shift work within an acute care hospital and effectiveness of: BP monitoring, increases in physical activity, positive nutritional changes, and the correlation between a primary care provider visits and lowering BP.

ELIGIBILITY:
Inclusion Criteria:

* Providence Health System's Southwest Washington Service Area (SWSA) employees
* Subjects who will be included in the intervention part of the study will have two consecutive BP readings of > 140/90
* Has or is willing to have collaborative PCP
* Understand and sign the informed consent form

Exclusion Criteria:

* Under the age of 18
* Has a severe systemic illness with life expectancy judged less than three years
* Has a severe vascular event such as Myocardial Infarction or Cerebral Vascular Event in the past 90 days
* Is enrolled in another therapeutic program or similar study, and
* Has a condition which, in the opinion of the investigators, may prevent the subject from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Reduction of blood pressure | 6 months
  The study will look for a reduction in blood pressure during a 6-month time frame among those identified at screening to have high blood pressure and who continue on in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Donahue, M.Ed., Principal Investigator — Providence Health and Services
Locations (1):
- Providence St. Peter Hospital, Olympia, Washington, United States